CLINICAL TRIAL: NCT00569101
Title: A Pilot Study for the Efficacy and Safety of Tacrolimus in the Treatment of Refractory Lupus Nephritis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Suhnggwon Kim, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-0706-049-211; 20070217867
Record Dates: First submitted 2007-12-04; First posted 2007-12-06 (Estimated); Last update posted 2007-12-06 (Estimated); Status verified 2007-12

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis | interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single (Experimental): single arm study (tacrolimus trial group)
  Interventions: Drug: tacrolimus

INTERVENTIONS:
Drug: tacrolimus — during the first 2 months : tacrolimus 0.1 mg/kg + prednisolone 0.8 mg/kg p.o. ,then after : tacrolimus 0.1 mg ~0.02 mg/kg + prednisolone tapering

SUMMARY:
The purpose of this protocol is to determine whether Tacrolimus and Prednisolone are effective and safe in the treatment of the cyclophosphamide-resistant, refractory diffuse proliferative lupus nephritis

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven lupus nephritis WHO Class IV , IV+V
* Previously treated by three times over of i.v. cyclophosphamide or 6 months more duration of immunosuppressive treatments (azathioprine, MMF, cyclophosphamide p.o.) for the lupus nephritis
* spot urine Protein creatinine raio > 1.0
* RBC > 5 /HPF on microscopic examination of urine

Exclusion Criteria:

* previous treatment of cyclosporine A or tacrolimus
* serum Creatinine lever : over 300 mmol/dl
* allergy to the macrolide antibiotics
* other systemic organ damage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2007-09; Study Completion 2008-03 (Estimated)

PRIMARY OUTCOMES:
Reducing proteinuria | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Suhnggwon Kim, MD, PhD, Principal Investigator — Korea : Seoul National University Hospital
Locations (1):
- SeoulNUH, Seoul, Chongno-gu, South Korea